CLINICAL TRIAL: NCT07131345
Title: A Single-Arm, Multicenter, Open-Label Phase Ib/II Clinical Study Exploring the Efficacy and Safety of Iparomlimab and Tuvonralimab Injection in Combination With Chemotherapy for the Treatment of Malignant Mesothelioma
Brief Title: Study of Iparomlimab and Tuvonralimab Plus Chemotherapy in Malignant Mesothelioma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Center, China (Other)
Collaborators: Qilu Pharmaceutical Co., Ltd. (Industry); Affiliated Cancer Hospital of Zhengzhou University (Unknown); Beijing Chest Hospital, Capital Medical University (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); Shaanxi Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Puyuan Xing, Department of Medical Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, National Cancer Center, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC5281
Record Dates: First submitted 2025-06-14; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Malignant Mesothelioma; Mesothelioma
Keywords: Malignant Mesothelioma; iparomlimab and tuvonralimab; immunotherapy
MeSH Terms: conditions — Mesothelioma, Malignant; Mesothelioma | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm: Iparomlimab and Tuvonralimab Combined with Chemotherapy (Experimental): Patients will receive Iparomlimab and Tuvonralimab (5 mg/kg) plus chemotherapy (pemetrexed and platinum drugs) every 3 weeks for 4-6 cycles, followed by maintenance therapy with Iparomlimab and Tuvonralimab for up to 2 years.
  Interventions: Drug: iparomlimab and tuvonralimab (Dual PD-1/CTLA-4 blockade) + chemotherapy

INTERVENTIONS:
Drug: iparomlimab and tuvonralimab (Dual PD-1/CTLA-4 blockade) + chemotherapy — Novel Bispecific Checkpoint Inhibition:
  QL1706(iparomlimab and Tuvonralimab) was generated by using MabPair, a new technological platform that enables the production of two antibodies close to their natural forms from a single host cell line and is manufactured as one product. QL1706 contains a mixture of anti-PD-1 IgG4 and anti-CTLA-4 IgG1 that were produced together in a fixed ratio. Each antibody was individually optimized to achieve desirable target coverage and antibody effector functions.
  Chemotherapy for first-line treatment (pemetrexed plus cisplatin or carboplatin )
  Chemotherapy for second-line treatment (pemetrexed, gemcitabine or vinorelbine)
  Other Names: QL1706+chemotherapy

SUMMARY:
This clinical trial aims to investigate the effectiveness and safety of a new treatment combination-Iparomlimab and Tuvonralimab (QL1706, a dual-function antibody targeting PD-1 and CTLA-4) combined with chemotherapy-for patients with malignant mesothelioma (MM). MM is a rare and aggressive cancer often linked to asbestos exposure. Current treatments have limited success, and this study seeks to explore a potentially more effective and safer option.

Study Design:

Phase Ib (Safety Phase): 6 patients will receive the combination therapy to assess safety. If no major safety issues arise, the study will proceed to Phase II.

Phase II (Efficacy Phase): 49 patients will be enrolled to evaluate treatment effectiveness. The study includes two groups for first-line treatment and second-line treatment.

DETAILED DESCRIPTION:
Study Rationale Malignant mesothelioma (MM) is a rare and aggressive cancer primarily associated with asbestos exposure. Despite advances in treatment, the prognosis remains poor, with a median overall survival (OS) of approximately 12-18 months for advanced disease. Current standard therapies include platinum-based chemotherapy combined with pemetrexed, immune checkpoint inhibitors (ICIs) such as nivolumab plus ipilimumab, or pembrolizumab with chemotherapy. However, these treatments have limitations, including significant toxicity (e.g., immune-related adverse events, irAEs) and modest survival benefits in certain populations.

The iparomlimab and tuvonralimab (QL1706) combination is a novel bispecific antibody therapy targeting PD-1 and CTLA-4, designed to enhance anti-tumor immune responses while minimizing toxicity. Preclinical and early clinical data suggest this dual checkpoint blockade may offer comparable efficacy to existing ICI combinations but with an improved safety profile. Given the unmet need for effective and tolerable therapies in MM, this study evaluates the clinical potential of iparomlimab and tuvonralimab combined with chemotherapy in Chinese patients.

Study Design

This is a single-arm, multicenter, open-label Ib/II trial with two sequential phases:

Phase Ib (Safety Run-In, n=6):

Evaluates the safety of iparomlimab and tuvonralimab + chemotherapy in patients with 1-3 prior lines of therapy.

Phase II (Expansion, n=49):

First-line cohort (n=39): Patients receive iparomlimab and tuvonralimab + pemetrexed/platinum (Simon two-stage design).

Second-line cohort (n=10): Fixed-sample evaluation of iparomlimab and tuvonralimab + investigator-selected chemotherapy.

Treatment Regimen

Induction Phase (4-6 cycles, Q3W):

Iparomlimab and tuvonralimab (5 mg/kg IV, Day 1)

Chemotherapy backbone:

First-line: Pemetrexed (500 mg/m²) + cisplatin (75 mg/m²) or carboplatin (AUC 5).

Second-line: Investigator's choice (pemetrexed, gemcitabine, or vinorelbine).

Maintenance Phase (up to 2 years, Q3W):

Iparomlimab and tuvonralimab monotherapy (5 mg/kg) until progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide informed consent prior to initiating any study-specific procedures.
* Male or female subjects aged ≥18 and ≤75 years.
* Histologically/cytologically confirmed malignant mesothelioma (MM), including malignant pleural mesothelioma (PM) and malignant peritoneal mesothelioma (PeM).
* Subjects with MM unsuitable for radical resection and/or radiotherapy per AJCC 8th Edition.
* Subjects who received neoadjuvant/adjuvant chemotherapy for radical surgery completed >6 months prior to current recurrent disease diagnosis, not counted in subsequent treatment lines.
* Prior systemic anti-tumor therapy requirements:

  * Safety run-in phase: ≥1 prior anti-tumor therapy line (maximum 3 lines)
  * Phase II first-line cohort: No prior systemic anti-tumor therapy
  * Phase II second-line cohort: Only 1 prior systemic anti-tumor therapy line
* ECOG performance status 0-2.
* Investigator-assessed life expectancy >3 months.
* Adequate hematological parameters.

Exclusion Criteria:

* Prior CTLA-4 inhibitors prohibited; prior PD-1/PD-L1 allowed unless discontinued for immune toxicity
* Immunomodulators within 14 days (e.g., thymosin, interleukin-2, interferon)
* Significant cardiovascular history within 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
ORR | From enrollment to the end of treatment at 8 weeks
  Objective Response Rate，Proportion of participants achieving complete response (CR) or partial response (PR) per modified RECIST 1.1 for mesothelioma

CONTACTS AND LOCATIONS:
Overall Officials: Puyuan Xing, MD, Principal Investigator — National Cancer Center, China

IPD SHARING:
Plan to Share IPD: No